CLINICAL TRIAL: NCT05106569
Title: Home-Based Spirometry Through Telemedicine in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Telespirometry in Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Eufrosina I. Young, Principal Investigator, State University of New York - Upstate Medical University
Other Study IDs: 1660190
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Pulmonary Function Test; Amyotrophic Lateral Sclerosis; Slow Vital Capacity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Spirometry; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SUNY Upstate: One of 2 ALS certified treatment centers in USA expected to recruit 50 subjects.
  Interventions: Diagnostic Test: Spirometry
- Atrium Health: One of 2 ALS certified treatment centers in USA expected to recruit 50 subjects.
  Interventions: Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Spirometry — All study participants will undergo pulmonary function testing using conventional spirometry in clinic and portable spirometry in clinic and at home. In-clinic conventional laboratory spirometry is compared with portable spirometry and Slow vital capacity is obtained in upright and supine positions.
  Other Names: Pulmonary Function Test

SUMMARY:
The investigators seek to validate Slow Vital Capacity (SVC) measurement in seated and supine positions using conventional and portable spirometry.

DETAILED DESCRIPTION:
SVC is obtained with in-clinic conventional spirometry, in-clinic portable spirometry, and in-home portable spirometry with respiratory therapist-supervised remote pulmonary function testing every two weeks in a six month prospective study of participants with a diagnosis of Amyotrophic Lateral Sclerosis. SVC decline over time, seated and supine, will be tracked with assessments for treatment changes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ALS as Clinically Possible, Clinically Probable, Laboratory-supported Probable and Clinically Definite ALS
2. 18 years old to 100 years old, English-speaking ALS subjects, male and female

Exclusion Criteria:

1. Use of non-invasive ventilation more than 16 hours daily
2. Non-English Speaker
3. Psychosis or severe mental illness
4. Use of high-dose sedating psychotropic medications determined to potentially interfere with task performance
5. Infection Control issues and specific Pulmonary, Cardiac, Vascular contraindications as listed in the Standardization of Spirometry 2019 Update (Graham 2019)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are invited to volunteer and recruited from ALS specialty care outpatient clinics at SUNY Upstate and Atrium Health.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ALS Functional Rating Scale, Revised (ALS FRSR) | 2 week intervals for 6 months
  Minimum 0, Maximum 48; Lower scores worse
Change from baseline SVC percent predicted at clinic | 3 months
  SVC measured at clinic in seated and supine positions using conventional and portable spirometer
Change from baseline SVC percent predicted at clinic | 6 months
  SVC measured at clinic in seated and supine positions using conventional and portable spirometer
Change from baseline SVC percent predicted at home | 2 week intervals for 6 months
  SVC measured from home in seated and supine positions using portable spirometer
Change from baseline Dyspnea in Amyotrophic Lateral Sclerosis 15 (DALS-15) | 2 week intervals for 6 months
  Minimum 0, Maximum 30; Higher scores worse
Change from baseline Hospital Anxiety and Depression Scale (HADS) | 6 months
  Minimum 0, Maximum 42; Higher scores worse
Change from baseline Amyotrophic Lateral Sclerosis Assessment Questionnaire-5 (ALSAQ-5) at 6 months | 6 months
  Minimum 0, Maximum 20; Higher scores worse
Change from baseline Amyotrophic Lateral Sclerosis Cognitive Behavioral Screen (ALS-CBCS) | 6 months
  Minimum 0, Maximum 20; Lower scores worse
Change from baseline Amyotrophic Lateral Sclerosis Cognitive Behavioral Screen (ALS-CBCS) ALS Caregiver Behavioral Questionnaire at 6 months | 6 months
  Minimum 0, Maximum 45; Lower scores worse
Change from baseline Amyotrophic Lateral Sclerosis Treatment Questionnaire | 2 week intervals for 6 months
  Reports usage of non-invasive ventilation, gastrostomy tube, ALS medications and ALS devices

CONTACTS AND LOCATIONS:
Overall Officials: Eufrosina Young, MD, Principal Investigator — SUNY Upstate
Locations (2):
- United States (2):
  - SUNY Upstate, Syracuse, New York
  - Atrium Health, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share Individual Patient Data collected during the study to research team from both sites.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years.
Access Criteria: Research team includes Principal investigators, sub-investigators, clinical research coordinators and respiratory therapists at each site, Pulmonologist Central Readers at SUNY Upstate. Deidentified data is shared with study sponsor MTPA.

REFERENCES:
- [Background] Geronimo A, Simmons Z. Evaluation of remote pulmonary function testing in motor neuron disease. Amyotroph Lateral Scler Frontotemporal Degener. 2019 Aug;20(5-6):348-355. doi: 10.1080/21678421.2019.1587633. Epub 2019 Apr 7. PMID 30957547
- [Background] Hegewald MJ, Gallo HM, Wilson EL. Accuracy and Quality of Spirometry in Primary Care Offices. Ann Am Thorac Soc. 2016 Dec;13(12):2119-2124. doi: 10.1513/AnnalsATS.201605-418OC. PMID 27598295
- [Background] Couratier P, Vincent F, Torny F, Lacoste M, Melloni B, Lemaire F, Antonini MT. Spirometer-dependence of vital capacity in ALS: validation of a portable device in 52 patients. Amyotroph Lateral Scler Other Motor Neuron Disord. 2005 Dec;6(4):239-45. doi: 10.1080/14660820510043244. PMID 16319028
- [Background] Masa JF, Gonzalez MT, Pereira R, Mota M, Riesco JA, Corral J, Zamorano J, Rubio M, Teran J, Farre R. Validity of spirometry performed online. Eur Respir J. 2011 Apr;37(4):911-8. doi: 10.1183/09031936.00011510. Epub 2010 Jul 22. PMID 20650985
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Result] Rutkove SB, Qi K, Shelton K, Liss J, Berisha V, Shefner JM. ALS longitudinal studies with frequent data collection at home: study design and baseline data. Amyotroph Lateral Scler Frontotemporal Degener. 2019 Feb;20(1-2):61-67. doi: 10.1080/21678421.2018.1541095. Epub 2018 Nov 28. PMID 30486680